CLINICAL TRIAL: NCT07258836
Title: A Phase 1, Open-Label Study to Evaluate the Safety, Biodistribution, Imaging Characteristics, and Radiation Dosimetry of [18F]LY4214835 in Healthy Volunteers and Participants With Cancer
Brief Title: A Study of [18F]LY4214835 in Healthy Volunteers and Participants With Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 27782; J6J-AV-AVCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms; Healthy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY4214835 (Cohorts 1 and 2) (Experimental): LY4214835 administered intravenously (IV)
  Interventions: Drug: LY4214835

INTERVENTIONS:
Drug: LY4214835 — Administered IV

SUMMARY:
The purpose of the study is to check how safe and well-tolerated [18F]LY4214835 injection is in healthy participants and participants with cancer. The study drug will be administered intravenously (IV) (into a vein). Participation in the study will last approximately 35 days.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1

  * Have a radiologically, cytologically, or histologically confirmed diagnosis of cancer
  * Are treatment-naïve to a systemic cancer therapy, OR have a documented disease progression on standard-of-care treatment (for example, failure of chemotherapy, targeted therapy or immunotherapy)
  * Have at least 1 imageable tumor that is 15 millimeter (mm) or larger in the longest diameter
* Cohort 2

  * Are overtly healthy at the Screening Visit and upon reporting to the clinic for the positron emission tomography (PET) Imaging Visit, as determined by medical evaluation including updated medical history, vital signs, physical examination, laboratory tests, and electrocardiogram (ECG)

Exclusion Criteria:

* Are pregnant or intend to become pregnant during their participation in the study
* Are breastfeeding or intending to breastfeed during their participation in the study
* Have a history of risk factors for Torsades de Pointes (for example, heart failure, hypokalemia, family history of Long QT Syndrome)
* Are actively receiving cancer therapy or are in between cycles of treatment
* Have a marked baseline prolongation of QT/corrected QT interval (QTc) interval (for example, repeated demonstration of a QTc interval greater than (>) 450 millisecond (ms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of Incidence of Adverse Events (AEs) | Baseline Through Day 3
  Evaluation of AEs regardless of causality, will be reported in the Reported AEs module
Number of Radiation Absorbed Dose Estimates in Body Organs to Obtain Whole-body Effective Dose | Baseline Through Day 3
  Determination of the radiation dosimetry absorbed dose in body organs and whole-body effective dose

SECONDARY OUTCOMES:
Number of Uptake of [18F]LY4214835 in Tumor Foci and Other Organs | Baseline Through Day 3
  Evaluation of the uptake of [18F]LY4214835 in tumor foci and other organs

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - Invicro, New Haven, Connecticut
  - Boston Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital (MGH), Charlestown, Massachusetts
  - BAMF Health Inc., Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ichor Research, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No